CLINICAL TRIAL: NCT03929796
Title: Evaluation of Prehospital Emergency Intubations Using Videolaryngoscopes
Brief Title: Video Analysis of Prehospital Emergency Intubations
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-02104
Record Dates: First submitted 2019-04-17; First posted 2019-04-29 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Intubation; Prehospital; Videolaryngoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Investigators' knowledge about pre-hospital emergency intubations is still limited. Various factors such as the average and the normal range of intubation time are still unknown. Since its launch Rega videotapes all intubation attempts with the C-MAC videolaryngoscope. The investigators prospectively analysed all routinely recorded intubation videos during one year performed by the Rega crews. The investigators analysed different parameters such as first pass success rate and the time to successfully intubate alongside with others. The goal was to find out more about this difficult procedure, about the problems which regularly occur and on what should be put particular emphasis during training.

DETAILED DESCRIPTION:
Pre-hospital emergency intubations are especially hazardous. The incidence of unanticipated difficult airways is higher (9,3 % of prehospital intubations are more difficult than anticipated). The first attempt intubation success rates are lower and the rate of complications compared to in-hospital emergency intubations is higher.

There is conflicting evidence if first attempt intubation success rate in prehospital intubations differs between intubations performed by videolaryngoscopy and direct laryngoscopy. On the other hand in pre-hospital airway management, the use of a C-MAC videolaryngoscope improved the visualization of glottic structures significantly.

The C-MAC has recently launched a new version, which allows videotaping of intubations. Rega decided to videotape all intubation attempts for legal purposes and quality control. These videos are stored at a Rega-based secure central database.

The Investigators knowledge there is only one video-enhanced retrospective analyses of a limited number of videolaryngoscopic pre-hospital intubations.

So far, there is no video-enhanced prospective analysis of first attempt intubation success rates or of the time necessary for successful intubation with videolaryngoscopes in the pre-hospital setting available. Therefore, the investigators intend to determine the exact first attempt intubation success rate and the time necessary to successfully intubate, alongside with parameters such as the Cormack/Lehane grade, blade position (Macintosh vs Miller) and others (e.g. difficulties during intubation) in the pre-hospital physician-staffed HEMS-setting. The investigators' goal is to learn more about what is actually happening during prehospital intubations and what type of difficulties may occur.

The investigators therefore prospectively analysed all routinely recorded intubation videos (using the built-in camera of the C-MAC videolaryngoscope) during one year performed by the Rega crews. These videos show real life intubations through the video function included in the device, only the image from the tip of the laryngoscopy blade inside the patient's mouth is recorded. The operating physicians additionally provided anonymous information about intubation management for each video after returning to the helicopter base

ELIGIBILITY:
Inclusion Criteria:

• All videos routinely taken from intubations performed during 1 year at the Swiss Air Rescue (Rega) at all 13 helicopter bases

Exclusion Criteria:

* Patients who were intubated primarily using other devices without a camera
* Intubations that were not recorded (missing data).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Patients which underwent Intubation performed by the Rega during 1year (15.02.18-14.02.19) because of medical or Trauma associated reasons (with or without cardiac arrest).
Sampling Method: Non-Probability Sample
Enrollment: 422 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
First attempt intubation success rate | Starts when the videolaryngoscope is inserted in the patients mouth for the first time and ends when the airway is secured
  Rate of a successful intubation at first attempt

SECONDARY OUTCOMES:
Overall success rate | Starts when the videolaryngoscope is inserted in the patients mouth for the first time and ends when the airway is secured
  The overall rate of successful intubation
Time intervals during intubation | Starts when the videolaryngoscope is inserted in the patients mouth for the first time and ends when the airway is secured
  entry-to-tube time (C-MAC crossing the lips to first appearance of tracheal tube in the field of view), time to intubation (C-MAC crossing the lips for the first time until passage of the tube through the vocal cords, the video is kept running throughout the intubation procedure), time between passage of the tube until removal of the blade from the mouth, overall time (from C-MAC crossing the lips for the first time until removal, the video is kept running throughout the intubation procedure), tube time (time from first appearance of the tube in the field until passage of the tube through the vocal cords), intubation time of the successful intubation attempt (C-MAC crossing the lips in the successful attempt until passage of the tube through vocal cords)
Number of intubation attempts | Starts when the videolaryngoscope is inserted in the patients mouth for the first time and ends when the airway is secured
  The total number of attempts needed for the intubation
Best C/L(Cormack/ Lehane 1-4) grade and best POGO (percent of glottis Opening 0 - 100 %) score | Starts when the videolaryngoscope is inserted in the patients mouth for the first time and ends when the airway is secured
  The best C/L and best POGO score achieved during the intubation
Additional Airway devices used | Starts when the videolaryngoscope is inserted in the patients mouth for the first time and ends when the airway is secured
  If additional devices have been used (e.g. Frova-like,catheter, Magill forceps, suction catheter)
Number of glottic hits | Starts when the videolaryngoscope is inserted in the patients mouth for the first time and ends when the airway is secured
  Number of attempts to advance the tracheal tube, but only glottic structures are being hit
Blade positioning | Starts when the videolaryngoscope is inserted in the patients mouth for the first time and ends when the airway is secured
  Blade positioning during intubation (Macintosh vs. Miller)
Unintended blade positions | Starts when the videolaryngoscope is inserted in the patients mouth for the first time and ends when the airway is secured
  Unintended blade positions (too deep, downfolding of epiglottis)
Secretion in the mouth and difficulties in visualisation because of it | Starts when the videolaryngoscope is inserted in the patients mouth for the first time and ends when the airway is secured
  Vomit, blood, saliva
Fogging of the camera | Starts when the videolaryngoscope is inserted in the patients mouth for the first time and ends when the airway is secured
  videolaryngoscope camera clear or fog
Oesophageal intubation | Starts when the videolaryngoscope is inserted in the patients mouth for the first time and ends when the airway is secured
  Oesophageal fail intubation during the procedure
Injury of the pharyngeal mucose due to the blade | Starts when the videolaryngoscope is inserted in the patients mouth for the first time and ends when the airway is secured
  Videolaryngoscope injury of the pharyngeal mucose due to the blade
Open or Closed vocal cords | Starts when the videolaryngoscope is inserted in the patients mouth for the first time and ends when the airway is secured
  Positioning of vocal cords if visible (open, closed), start of movement of vocal cords

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Theiler, Prof., Principal Investigator — Department of Anaesthesiology and Pain Therapy, Bern University Hospital
Locations (1):
- Bern University Hospital and University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hossfeld B, Frey K, Doerges V, Lampl L, Helm M. Improvement in glottic visualisation by using the C-MAC PM video laryngoscope as a first-line device for out-of-hospital emergency tracheal intubation: An observational study. Eur J Anaesthesiol. 2015 Jun;32(6):425-31. doi: 10.1097/EJA.0000000000000249. PMID 25886716
- [Background] Carlson JN, Quintero J, Guyette FX, Callaway CW, Menegazzi JJ. Variables associated with successful intubation attempts using video laryngoscopy: a preliminary report in a helicopter emergency medical service. Prehosp Emerg Care. 2012 Apr-Jun;16(2):293-8. doi: 10.3109/10903127.2011.640764. Epub 2011 Dec 22. PMID 22191806
- [Background] Kim SY, Park SO, Kim JW, Sung J, Lee KR, Lee YH, Hong DY, Baek KJ. How much experience do rescuers require to achieve successful tracheal intubation during cardiopulmonary resuscitation? Resuscitation. 2018 Dec;133:187-192. doi: 10.1016/j.resuscitation.2018.08.032. Epub 2018 Aug 30. PMID 30172693
- [Background] Gunning M, O'Loughlin E, Fletcher M, Crilly J, Hooper M, Ellis DY. Emergency intubation: a prospective multicentre descriptive audit in an Australian helicopter emergency medical service. Emerg Med J. 2009 Jan;26(1):65-9. doi: 10.1136/emj.2008.059345. PMID 19104110
- [Background] Smith CM, Yeung J. Airway management in cardiac arrest-Not a question of choice but of quality? Resuscitation. 2018 Dec;133:A5-A6. doi: 10.1016/j.resuscitation.2018.10.009. Epub 2018 Oct 15. No abstract available. PMID 30336234